CLINICAL TRIAL: NCT06820411
Title: Y-SCOPE Study: a Pilot Study to Assess Optimal Prevention and Outcome Improvement in Young Ischemic Stroke
Brief Title: A Pilot Study to Assess Optimal Prevention and Outcome Improvement in Young Ischemic Stroke
Acronym: Y-SCOPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Y-SCOPE Study; Neuro Virtual Hospital (Other Grant/Funding Number: POR-FERS REGIONE LOMBARDIA 2014-2020)
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Ischemic Stroke At a Young Age; Secondary Prevention
Keywords: Young stroke prevention; Ischemic Stroke in Young Adults; Secondary Stroke Prevention; Lifestyle Modification After Stroke; Wearable Health Monitoring in Stroke; Stroke Risk Factor Management; Pilot Study in Stroke Prevention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Young Stroke Clinic Intervention (Experimental): Participants in this arm will receive specialized care at the Young Stroke Clinic, designed for individuals aged 18-65 who have experienced an ischemic stroke or high-risk TIA. The intervention includes:
  Personalized risk factor management, focusing on blood pressure, cholesterol, smoking cessation, diet, and physical activity.
  Intensive lifestyle counseling to encourage adherence to secondary prevention strategies.
  Use of a wearable device (Whoop 4.0) to monitor heart rate variability, sleep patterns, and physical activity.
  Regular follow-up visits with neurologists to track progress and provide guidance.
  The goal is to optimize cardiovascular health, reduce recurrent stroke risk, and enhance long-term outcomes.
  Interventions: Behavioral: Young Stroke Clinic Lifestyle Intervention; Other: Standard Post-Stroke Care
- Standard Care Control Group (Active Comparator): Participants in this arm will receive standard post-stroke care based on current clinical guidelines. This includes:
  Routine follow-up visits with healthcare providers. Medical management of stroke risk factors such as hypertension, diabetes, and dyslipidemia.
  General lifestyle recommendations, including advice on diet, physical activity, and smoking cessation, as provided in standard clinical practice.
  Unlike the experimental group, this arm does not include structured intensive lifestyle counseling, dedicated stroke clinic follow-ups, or wearable device monitoring.
  Interventions: Other: Standard Post-Stroke Care

INTERVENTIONS:
Behavioral: Young Stroke Clinic Lifestyle Intervention — The Young Stroke Clinic Lifestyle Intervention is a structured program designed for young adults (18-65 years) recovering from ischemic stroke or high-risk TIA. It includes:
  * Personalized risk factor management targeting blood pressure, cholesterol, smoking cessation, and lifestyle habits.
  * Intensive lifestyle counseling to improve diet, physical activity, and overall cardiovascular health.
  * Wearable device monitoring (Whoop 4.0) to track heart rate variability, sleep patterns, and physical activity.
  * Regular follow-up visits at a dedicated stroke clinic with tailored guidance from neurologists.
  Arms: Young Stroke Clinic Intervention
Other: Standard Post-Stroke Care — The Standard Post-Stroke Care group will receive usual medical management based on current clinical guidelines for secondary stroke prevention. This includes:
  * Routine follow-up visits with healthcare providers.
  * Standard medical treatment for stroke risk factors (e.g., blood pressure, cholesterol, diabetes).
  * General lifestyle recommendations on diet, physical activity, and smoking cessation as part of routine clinical care.

SUMMARY:
Purpose The Y-SCOPE study aims to improve the health and recovery of young adults aged 18 to 65 who have experienced an ischemic stroke or a high-risk transient ischemic attack (TIA). By focusing on personalized care and lifestyle changes, the study seeks to reduce the chances of another stroke and promote better long-term health.

Background While strokes are often associated with older adults, recent studies have shown an increase in ischemic strokes among younger individuals. Given that younger patients are typically in their working years and have longer life expectancies, a stroke can lead to significant long-term disability and economic challenges. Addressing the unique needs of this population is crucial for effective care and research.

Study Design

This is an open-label pilot study, meaning both participants and researchers know which treatments are being administered. The study will enroll 36 participants who will be randomly assigned in a 2:1 ratio:

Intervention Group (24 participants): Will receive personalized care through a dedicated "Young Stroke Clinic." Control Group (12 participants): Will receive standard post-stroke care.

Intervention Details

Participants in the intervention group will:

* Attend specialized clinic visits focused on young stroke patients.
* Receive intensive counseling to manage risk factors such as high blood pressure, cholesterol, and lifestyle habits.
* Be provided with a wearable device (Whoop 4.0) to monitor health metrics like heart rate, sleep patterns, and physical activity.

Duration The study will last for 12 months, with an 8-month enrollment period and a minimum follow-up of 6 months for each participant.

Eligibility Criteria

Inclusion:

* Ages 18 to 65.
* Diagnosed with acute ischemic stroke or high-risk TIA.
* Moderate to low cardiovascular health status.
* Able to perform daily activities independently or with minimal assistance.

Exclusion:

* Pregnancy.
* Lack of access to a compatible smartphone for device monitoring.
* Inability to commit to the follow-up schedule.

Objectives

* Primary Objective: Assess the feasibility of the study by evaluating participant eligibility, consent rates, adherence to interventions, and retention rates.
* Secondary Objectives: Compare health outcomes between the intervention and control groups, including:

Improvement in cardiovascular health scores. Reduction in major cardiovascular events. Enhancements in physical activity, diet, sleep quality, and smoking cessation. Changes in inflammatory markers in the blood.

Potential Benefits While this is a pilot study and may not provide definitive evidence of effectiveness, it aims to develop a tailored secondary prevention strategy for young stroke patients. The personalized approach could lead to better management of risk factors, improved quality of life, and a reduction in recurrent strokes and other cardiovascular events.

Participation Participants will be required to attend scheduled clinic visits, engage in counseling sessions, and use the provided wearable device consistently. Regular monitoring and feedback will be integral parts of the program.

Confidentiality All personal health information and data collected during the study will be kept confidential and used solely for research purposes.

This study is conducted by the Neurology Department and Stroke Unit at the IRCCS Mondino Foundation.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 65 years.
* Diagnosis: Acute ischemic stroke or high-risk transient ischemic attack (TIA) (ABCD2 score ≥ 6).
* Cardiovascular Health Status: Low or moderate cardiovascular health, assessed by the American Heart Association's Life's Essential 8 (LE8) Score.
* Functional Independence: Modified Rankin Scale (mRS) score of 0 to 2 at enrollment.
* Ability to Participate: Participants must be able to adhere to the study's follow-up visits and intervention requirements.

Exclusion Criteria:

* Pregnancy.
* Inability to Use Wearable Device: Participants must have a compatible smartphone for the wearable device (Whoop 4.0).
* Medical Conditions: Any condition that prevents participation in the follow-up program (e.g., severe cognitive impairment, terminal illness).
* Unwillingness to Participate: Individuals who decline consent or are unable to comply with study requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the Young Stroke Clinic Lifestyle Intervention | From baseline to study completion (12 months)
  The primary outcome assesses the feasibility of the intervention based on four key metrics:
  * Eligibility Rate: Proportion of eligible participants among all screened young stroke patients.
  * Consent Rate: Proportion of eligible patients who agree to participate.
  * Adherence Rate: Degree of compliance with lifestyle recommendations, assessed through validated scoring tools.
  * Dropout Rate: Proportion of participants who discontinue before study completion.
  These measures will determine whether the intervention is practical and acceptable for future large-scale trials.

SECONDARY OUTCOMES:
Impact of the Young Stroke Clinic Intervention on Cardiovascular Health and Lifestyle Factors | Baseline, 3 months, and 6 months
  The study evaluates the effect of the intervention on cardiovascular health and lifestyle modifications. Key measures include:
  * Cardiovascular Health Score (LE8): Comparison at baseline, 3 months, and 6 months.
  * Major Adverse Cardiovascular Events (MACE): Incidence of recurrent stroke, myocardial infarction, or cardiovascular death.
  * Physical Activity, Sleep, and Smoking Behavior: Assessed through validated questionnaires (International Physical Activity Questionnaire, Pittsburgh Sleep -Quality Index, 14-MEDAS, and daily cigarette count).
  * Wearable Device Metrics: Heart rate variability, resting heart rate, and sleep duration.
  * Inflammatory Biomarkers: Serum levels of TNF-alpha, IL-6, IL-10, and other cytokines.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS National Neurological Institute "C. Mondino" Foundation, Pavia, Pavia 27100, Pavia, PV, Italy

IPD SHARING:
Plan to Share IPD: No